CLINICAL TRIAL: NCT01440556
Title: Allogeneic Bone Marrow Transplantation From Unrelated Donors in Multiple Myeloma: a Study From the Italian Bone Marrow Transplantation Donor Registry
Brief Title: Allogeneic Bone Marrow Transplantation From Unrelated Donors in Multiple Myeloma
Acronym: MM2011
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Responsible Party: Principal Investigator, Benedetto Bruno, Dr, Azienda Ospedaliera San Giovanni Battista
Other Study IDs: IBMDR-MM-2011
Record Dates: First submitted 2011-09-23; First posted 2011-09-26 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Multiple Myeloma; Allogeneic Transplantation
Keywords: Allogeneic bone marrow transplantation; Multiple myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Autologous hematopoietic cell transplantation is currently considered the standard therapy of multiple myeloma (MM) for elegible patients. On the contrary, despite new developments in transplant procedures and supportive care, allogeneic bone marrow transplantation is less commonly used due to high transplant related mortality (TRM).

No consensus statement about allografting in MM has so far been reached and only a minority of patients undergoing allografting are enrolled in prospective clinical trials.

Moreover, use of unrelated donors is considerably increased over the time and the recent activity survey of European Group for Blood and Marrow Transplantation (EBMT) showed that the number of allografts from unrelated donor is higher than that one from HLA-identical siblings in Europe.

In order to evaluate trends in allograft from unrelated donors in multiple myeloma patients, the investigators plan to conduct a restrospective study through the Italian Bone Marrow Transplantation Registry (IBMDR) over a period ranging since 2000 to 2009. Data will be collected from the central data management system Promise (Project Manager Internet Server) used by EBMT and from IBMDR.

The aim of the study is to evaluate the role of unrelated donor allograft in multiple myeloma over the last decade and hopefully offer recommendations on patient selection. Primary endpoints of the study are: a) Overall Survival (OS) from diagnosis and from the allograft b) Event-Free-Survival (EFS) from the allograft. Disease response criteria will be defined according to the International Uniform Response Criteria for multiple myeloma. Transplant related mortality, Graft-Versus-Host-Disease (GVHD), either acute or chronic (limited/extensive) will be evaluated as cumulative incidences. Univariate and multivariate analysis will be calculated for the transplant-related and patient-related characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma patients treated with allogeneic bone marrow transplantation from unrelated donors (from 2000 to 2009: Centri Trapianto GITMO)

Exclusion Criteria:

* No exclusion criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple Myeloma patients
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 year
Event-free survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Benedetto Bruno, Dr, Principal Investigator — A.O.U.San Giovanni Battista di Torino
Locations (1):
- A.O.U.San Giovanni Battista di Torino, Torino, Italy